CLINICAL TRIAL: NCT05517876
Title: A Retrospective, Observational, Multicenter, Study to Collect Clinical Safety and Performance Data on POLYMAILLE®C
Status: Completed | Type: Observational
Sponsor: Perouse Medical (Industry)
Collaborators: Eclevar Medtech (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-PMC-01
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Abdominal Vascular Surgery; Peripheral Vascular Surgery; Vascular Prothesis; Aneurysm Abdominal; Aneurysm; Peripheral; Obliterative Arterail Disease
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vascular abdominal or peripheral surgery — replacement or bypass of arteries presenting aneurysm or obliterative arterial disease. Their indication is restricted to abdominal and peripheral surgery not crossing the knee flexion crease.
  Abdominal vascular surgery includes abdominal aorto-aortic and/or aorto-iliac and/or aorto-femoral vascular repair, i.e. graft implantation with proximal anastomosis to abdominal aorta (supra and/or infra-renal).
  Peripheral vascular surgery includes peripheral arteries repair, i.e. graft implantation with no aortic anastomosis, and/or extra-anatomic vascular repair such as axillo-femoral and/or crossover bypass (femoro-femoral and/or ilio-femoral).

SUMMARY:
Purpose of the study is to describe safety and performance of POLYMAILLE® C from a minimum of 200 subjects will be evaluated. A minimum of 100 subjects will be evaluated for each main location of surgery (abdominal and peripheral).

Follow-up At least 1 year follow-up after surgery until a maximum of 5 years. POLYMAILLE®C vascular prostheses are indicated for replacement or bypass of arteries presenting aneurysm or obliterative arterial disease. Their indication is restricted to abdominal and peripheral surgery not crossing the knee flexion crease.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all the following inclusion criteria in order to be eligible for inclusion in the study: Patient has a minimum of 1-year post-operative follow-up data available, or complete data to death

Exclusion Criteria:

* Patients who have objected to the collect of their data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All potential subjects and will select those who are appropriate for study inclusion, i.e. subjects implanted with POLYMAILLE® C for at least one year, or with complete data to death. As the study explores real world data, there is no exclusion criteria for subjects and all subjects with POLYMAILLE® C implanted for at least one year and up to 5 years will be included in the study.
  All data will be retrieved from medical charts for each patient from time of surgery (considered as index date) until a maximum of 5 years after surgery.
  A minimum of 100 subjects will be evaluated for each main location of surgery (peripheral and abdominal).
Sampling Method: Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Primary performance endpoint | 1 year
  primary patency rate
Primary safety endpoint | 30 days
  mortality rate

SECONDARY OUTCOMES:
Procedural success rate | 5 years
  * Ability to use with no need for replacement by another device and,
  * Effective vascular flow restoration after procedure and,
  * In case of aneurysm, exclusion of aneurysmal portion after procedure.
Primary patency rate | 5 years
  rate of patent grafts without any procedure or intervention of the conduit itself
Primary assisted patency rate | 5 years
  rate of patent grafts, with or without procedure or intervention of the conduit itself after device implantation, such as endovascular balloon angioplasty or anastomotic revision, however with graft never thrombosed (graft occlusion)
Secondary patency rate | 5 years
  rate of patent grafts, with or without procedure or intervention of the conduit itself after device implantation, such as endovascular balloon angioplasty or anastomotic revision, lysis and/or thrombectomy.
Device Failure | 5 years
  * Uncontrolled blood leakage from device
  * Loss of structural integrity, e.g. rupture and/or exaggerated dilation (> 50 %)
  * Occlusion of the device
  * Total or partial replacement of the device required
Mortality rate | 5 years
  freedom % from death
Limb salvage rate | 5 years
  freedom % from target limb amputation
Adverse events | 5 years
  any documented adverse events, including anticipated and non-anticipated adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes', Nantes, France

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT05517876/Prot_000.pdf